CLINICAL TRIAL: NCT02822950
Title: A Study of Avycaz (Ceftazidime/Avibactam) Pharmacokinetics/Pharmacodynamics (PK/PD) in Critically Ill Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Gary E. Stein, Pharm.D., Professor of Medicine, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIT-USA-000832
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Pharmacokinetics of Avycaz in ICU Patients
MeSH Terms: interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ceftazadime/avibactam (Other): Ceftazadime/avibactam 2500 mg (1250 mg for CrCl 31-50 mL/min) IV over 120 minutes, every 8 hours [other antibiotics can also be administered as needed]. Patients will receive at least 3 doses (steady-state) of Avycaz prior to obtaining serum samples.
  Interventions: Drug: Ceftazidime/avibactam

INTERVENTIONS:
Drug: Ceftazidime/avibactam — Ceftazadime/avibactam dosing in ICU patients
  Other Names: Avycaz

SUMMARY:
The purpose of this study is to analyze the PK/PD of AvyCaz in critically ill patients in the Intensive Care Unit (12). This study will include medical and post-surgical patients who develop an infection where Avycaz can be utilized. Since these patients will have variable PK parameters, the investigators will also analyze (time-kill) these serum concentrations (ex vivo) against relevant clinical isolates (e.g. GNR with ESBL or KPC) from the ICU to determine microbiologic activity of Avycaz in critically ill patients with variable characteristics. Monte-Carlo simulations will also be conducted against clinical ICU isolates (JMI labs) to help determine appropriate dosing schedules based upon these PK parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18y/o) patients with a medical or post-surgical infection such as skin/soft tissue infections, urinary infections, IA infections and pneumonia (including VAP)
* Patients requiring intensive care (critically ill patients) in the med/surg ICU (APACHE II score ≥ 15)
* Patients prescribed Avycaz for their infection will receive FDA recommended dosages and times of administration
* Written informed consent

Exclusion Criteria:

* Pregnant Patients, patients older than 90 y/o, those with CrCl < 30 mL/min, patients with a BMI > 45 Kg/m2, patients unable to provide serum samples, and those with the risk of imminent death during the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Stein, PharmD, Principal Investigator — Michigan State University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ceftazadime/Avibactam
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ceftazadime/Avibactam
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 55 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean (SD) Ceftazadime/Avibactam Pharmacokinetic (PK) Volume of Distribution Parameter in Intensive Care Patients
Time Frame: 2,4,6, 8 hours after receiving the drug
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ceftazadime/Avibactam
Number analyzed (Participants) | 10
Liter | 34 (12)

2. Primary Outcome: Mean (SD) Ceftazadime/Avibactam Pharmacokinetic Half Life Parameter in Intensive Care Patients
Time Frame: 2,4,6, 8 hours after receiving the drug
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ceftazadime/Avibactam
Number analyzed (Participants) | 10
Hours | 4.3 (1.9)

3. Primary Outcome: Mean (SD) Ceftazadime/Avibactam Pharmacokinetic Clearance of Drug Parameter in Intensive Care Patients
Time Frame: 2,4,6, 8 hours after receiving the drug
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Ceftazadime/Avibactam
Number analyzed (Participants) | 10
Liters/hour | 6.4 (3.4)

4. Primary Outcome: Mean (SD) Ceftazadime/Avibactam Pharmacokinetic Area Under Serum Curve (mg*h/L) Parameter in Intensive Care Patients
Time Frame: 2,4,6, 8 hours after receiving the drug
Measure: Mean (Standard Deviation); unit: mg*hour/liters
Arm/Group | Ceftazadime/Avibactam
Number analyzed (Participants) | 10
mg*hour/liters | 343 (47)

5. Primary Outcome: Mean (SD) Ceftazadime/Avibactam Pharmacokinetic (PK) Maximum Serum Concentration in Intensive Care Patients
Time Frame: 2,4,6, 8 hours after receiving the drug
Measure: Mean (Standard Deviation); unit: mg/liter
Arm/Group | Ceftazadime/Avibactam
Number analyzed (Participants) | 10
mg/liter | 48 (17)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Ceftazadime/Avibactam
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT02822950/Prot_SAP_000.pdf